CLINICAL TRIAL: NCT03121261
Title: The Effect of Local Anesthetic and Clonidine on the Cutaneous Silent Period During and After Spinal Anesthesia
Brief Title: The Effect of Local Anesthetic and Clonidine on the Cutaneous Silent Period During Spinal Anesthesia
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Sandra Graf Zupcic, Neurology Specialist, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 070219812014
Record Dates: First submitted 2017-04-11; First posted 2017-04-20 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Inguinal Hernia; Spinal Anesthesia
Keywords: levobupivacaine; nerve fibers; clonidine
MeSH Terms: conditions — Hernia, Inguinal | interventions — Levobupivacaine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.5% levobupivacaine with 0.015% clonidine (Experimental): 0.5% levobupivacaine 15 mg with 0.015% clonidine 50 mcg and 40% glucose 0.5 ml will be preformed as subarachnoid block
  Interventions: Drug: levobupivacaine; Drug: clonidine
- 0.5% levobupivacaine with 0.9% saline (Active Comparator): 0.5% levobupivacaine 15 mg with 0.33 ml of 0.9% saline and 40% glucose 0.5 ml will be preformed as subarachnoid block
  Interventions: Drug: levobupivacaine; Drug: clonidine

INTERVENTIONS:
Drug: levobupivacaine — Comparing: 0.5% levobupivacaine 15 milligrams (mg) , 0.015% clonidine 50 micrograms (mcg) and 40% glucose 0.5 milliliters (ml) with 0.5 levobupivacaine 15 mg , 0.9% saline 0.33 ml and 40% glucose 0.5 ml
  Other Names: chirocaine
Drug: clonidine — Comparing: 0.5% levobupivacaine 15 mg , 0.015% clonidine 50 mcg and 40% glucose 0.5 ml with 0.5 levobupivacaine 15 mg , 0.9% saline 0.33 ml and 40% glucose 0.5 ml
  Other Names: catapressan

SUMMARY:
The cutaneous silent period is a non-invasive technique that gives insight into the function of thin A delta fibers and as such can be a complement to conventional electrophysiological methods used to study the peripheral nerves. Clonidine is a selective partial agonist of the alpha-2 receptors which, added intrathecally to levobupivacaine, enhances the effect of a local anesthetic, prolongs sensory and motor block during local anesthesia and extends the length of post-operative analgesia. It is believed that clonidine achieves this effect by activating the postsynaptic alpha-2 receptors in the gelatine substance of the spinal cord and blocking the conduction of A-delta and C fibers. The aim of the study is to examine functional changes of Aδ - fibers during the application of spinal anesthesia by measuring the cutaneous slinet period and compare the effect of intrathecal administration of a combination of local anesthetic and clonidine in the quiet skin period in relation to the application of local anesthetic only.

ELIGIBILITY:
Inclusion Criteria:

ASA one and two status BMI 18,5 to 24

Exclusion Criteria:

Coagulation disorders Polyneuropathy Diabetes mellitus Alcoholism Systemic inflammatory and malignant diseases Stroke

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
4 Item Duration of Latency and duration of the cutaneous silent period | 24 hours perioperative
  Duration of latency and duration of the cutaneous silent (msec) period before subarahnoid block, after regression of motor block, sixth hour of intrathecal administration, 24 hours after intrathecal administration

SECONDARY OUTCOMES:
Duration of motor block | 24 hours perioperative
  The duration of motor block and its regression will be monitored by Bromage scale:0- Bromage patient can perform movements in the hip, knee and foot. Bromage 1-patient can not perform movements in the hip, but can flexes the knee and move the foot, Bromage 2- patient can not perform movements in the hip and knee, but can move a foot. Bromage 3- patient can not perform movements in the hip, knee nor move the foot. The time of intrathecal levobupivacaine solution or levobupivacaine and clonidine solution is considered to be time zero.
Duration of sensory block | 24 hours perioperative
  The time needed for the regression of sensory block in two dermatome will be measured; the time (min) required for a regression in the S1 dermatome, the time required to restore motor functions in Bromage 0 and the duration of analgesia(min).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Hospital Dubrava, Zagreb, Croatia

REFERENCES:
- [Background] Inghilleri M, Cruccu G, Argenta M, Polidori L, Manfredi M. Silent period in upper limb muscles after noxious cutaneous stimulation in man. Electroencephalogr Clin Neurophysiol. 1997 Apr;105(2):109-15. doi: 10.1016/s0924-980x(97)96579-6. PMID 9152203
- [Background] Mota IA, Fernandes JB, Cardoso MN, Sala-Blanch X, Kofler M, Valls-Sole J. Temporal profile of the effects of regional anesthesia on the cutaneous reflexes of foot muscles. Exp Brain Res. 2015 Sep;233(9):2587-96. doi: 10.1007/s00221-015-4329-2. Epub 2015 May 30. PMID 26025613
- [Result] Uncini A, Kujirai T, Gluck B, Pullman S. Silent period induced by cutaneous stimulation. Electroencephalogr Clin Neurophysiol. 1991 Oct;81(5):344-52. doi: 10.1016/0168-5597(91)90023-q. PMID 1718720